CLINICAL TRIAL: NCT03561415
Title: Universal Posaconazole Prophylaxis Versus Pre-emptive Posaconazole Therapy for Fungal Infection Management Post-lung Transplantation
Brief Title: Universal Prophylaxis Versus Pre-emptive Therapy With Posaconazole Post-Lung Transplant
Acronym: UPPRITE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Bayside Health (Other Government)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 204/17
Record Dates: First submitted 2018-05-09; First posted 2018-06-19 (Actual); Last update posted 2018-06-19 (Actual); Status verified 2018-06

CONDITIONS: Fungal Infection
Keywords: Lung transplant, prophylaxis, pre-emptive
MeSH Terms: conditions — Mycoses

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Universal posaconazole prophylaxis (Experimental): Universal posaconazole prophylaxis: All patients will start posaconazole modified release tablet (300mg daily ) between Day 4 and Day 14 post lung or heart-lung transplantation for 3 months.
  Interventions: Other: Universal Posaconazole Prophylaxis
- Pre-emptive posaconazole therapy (Experimental): Pre-emptive posaconazole therapy: Posaconazole will be started if a fungal pathogen is identified or there is serological evidence of a fungal pathogen in the absence of any evidence of invasive fungal disease and given for 3 months.
  Interventions: Other: Pre-emptive Posaconazole Therapy

INTERVENTIONS:
Other: Universal Posaconazole Prophylaxis — All patients assigned to this arm will start posaconazole between Day 4 and Day 14 post lung or heart-lung transplant for a minimum of 3 months.
  Arms: Universal posaconazole prophylaxis
Other: Pre-emptive Posaconazole Therapy — Posaconazole will be started if a fungal pathogen is identified or there is serological evidence of a fungal pathogen in the absence of any evidence of invasive fungal disease for 3 months.
  Arms: Pre-emptive posaconazole therapy

SUMMARY:
This trial will examine 2 ways of using the antifungal posaconazole to prevent invasive fungal disease and the precipitation of chronic rejection post lung transplantation.

DETAILED DESCRIPTION:
Lung transplantation (LT) is an increasingly used treatment for end-stage respiratory disease. However, it is expensive, with hospital costs alone estimated at >US$500,000/transplant. Fungal infection and chronic lung allograft dysfunction (CLAD) are the major complications of LT. They pose the greatest threat to long-term survival and are reported to occur in 12-50% of LT recipients and cause death in 21.7-82% of these.

Fungal infections occur in 3 major forms in LT recipients, namely colonisation, trachea-bronchial disease and invasive (or end-organ) disease. Whilst invasive fungal disease (IFD) is associated with the highest mortality, colonisation poses the greatest clinical challenge. It is the most common manifestation, can progress to IFD and can precipitate CLAD. Antifungal prophylaxis is used to minimise the risks associated with colonisation.

Two main antifungal prophylaxis strategies are used. Universal prophylaxis (UP) is defined as the administration of antifungal agents to all patients post-LT. Most centres use UP. A systematic review and meta-analysis showed neither Aspergillus colonisation nor invasive aspergillosis (IA) (the commonest fungal infection in LT recipients) were reduced by UP. Yet it caused side-effects in 29.6%.

The pre-emptive strategy is defined as the administration of antifungal agents when a fungal pathogen (including in donor specimens) is detected or there is serological evidence of a fungal pathogen in the absence of IFD from a post-LT surveillance bronchoscopy or other clinical investigations (i.e. colonisation).Observational data suggest that a pre-emptive strategy has similar IA incidence rates but fewer adverse drug reactions (ADR) than UP (16.1%). It has been estimated that a pre-emptive strategy can reduce antifungal drug use by 43%.

No direct comparison of the efficacy, safety and cost of the two strategies has been performed to date. Thus, a randomised controlled trial (RCT) is needed to determine the optimal strategy to reduce the impact of fungal infection in LT recipients. However, before we embark on a definitive phase III RCT powered for clinical outcomes we will perform a pilot feasibility RCT to generate data and answer practical questions to better inform the design of the definitive phase III RCT powered for clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female aged ≥ 18 years
2. Undergoing bilateral sequential lung transplant (BSLT) or heart-lung transplant (HLT) including re-do transplant
3. Able to give written informed consent
4. Able to understand and comply with all trial requirements

Exclusion Criteria:

1. Less than 18 years of age
2. Scheduled to undergo a single-lung transplant (known risk factor for IFD)
3. Scheduled to undergo multi-organ transplant, other than HLT
4. Recipients who will not be followed up for 1-year post-transplant at one of the trial sites
5. Isolation of a mould within the 12 months prior to screening
6. Evidence of a mycetoma within the 12 months prior to screening
7. Proven or probable IFD within the 12 months prior to screening
8. Patients with moderate or severe liver disease as defined by aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 5 times the upper limit of normal (ULN)
9. Any other severe condition which in the site investigator's judgement may interfere with the trial evaluations or severely affect the patients safety
10. Previous inclusion in the trial
11. Currently enrolled in an antifungal or other investigational drug trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2018-07-02 (Estimated); Primary Completion 2020-09-30 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
Composite of: screened that are eligible, eligible that are enrolled, lost to follow-up or are withdrawn from the trial, receive their allocated treatment throughout the trial participation and have missing data during trial data collection. | 2 years and 3 months
  Feasibility outcome

SECONDARY OUTCOMES:
Composite of: at least one episode of fungal pneumonia, fungal tracheobronchitis, or bronchial anastomotic fungal infection; diagnosed as having CLAD or died regardless of cause | 2 years and 3 months
  Efficacy outcome
Fungal pneumonia, fungal tracheobronchitis, or bronchial anastomotic fungal infection rates | 2 years and 3 months
  Efficacy outcome
CLAD rates | 2 years and 3 months
  Efficacy outcome
All-cause mortality rates | 2 years and 3 months
  Efficacy outcome
Fungal pneumonia, fungal tracheobronchitis, or bronchial anastomotic fungal infection-related mortality rates | 2 years and 3 months
  Efficacy outcome
CLAD-related mortality rates | 2 years and 3 months
  Efficacy outcome
Time to development of fungal pneumonia, fungal tracheobronchitis, bronchial anastomotic fungal infection | 2 years and 3 months
  Efficacy outcome
Time to diagnosis of CLAD | 2 years and 3 months
  Efficacy outcome
Costs associated with allocated arm including number of hospital admissions | 2 years and 3 months
  Efficacy outcome
Quality of life (QoL) using Short Form Survey (sf-36) to measure patient health | 2 years and 3 months
  Efficacy outcome
Acute rejection rates | 2 years and 3 months
  Safety outcome
Posaconazole adverse drug reaction (ADR) rates | 2 years and 3 months
  Safety outcome
Proportion of patients who discontinue posaconazole because of an ADR | 2 years and 3 months
  Safety outcome
Total duration on posaconazole | 2 years and 3 months
  Safety outcome

CONTACTS AND LOCATIONS:
Overall Officials: Orla Morrissey, Study Chair — The Alfred
Locations (3):
- Australia (3):
  - St. Vincent's Hospital, Sydney, New South Wales
  - The Prince Charles Hospital, Brisbane, Queensland
  - Alfred Health, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: No